CLINICAL TRIAL: NCT05339217
Title: Efficacy and Immunological Evaluation of Telitacicept and Low Dose IL2 in the Treatment of Systemic Lupus Erythematosus: a Randomise Prospective Study
Brief Title: Efficacy and Immunological Evaluation of Telitacicept and Low Dose IL2 in the Treatment of Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liu Tian (Other)
Responsible Party: Sponsor-Investigator, Liu Tian, associate professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peking2022SLE
Record Dates: First submitted 2022-04-02; First posted 2022-04-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Telitacicept; IL-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept; RC-18; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telitacicept and low dose IL2 (Experimental): 160mg Telitacicept was subcutaneously injected to patients with systemic lupus erythematosus at the outer side of upper arm every week for 24 weeks.
  Interleukine-2 was first added to the original treatment for systemic lupus erythematosus with 1 million IU qod for 12 weeks, injected subcutaneously at the outer side of upper arm, abdomen and thigh, then the same dose of IL2 was injected once a week for 12 weeks subcutaneously.
  Interventions: Drug: Telitacicept; Drug: Interleukin-2
- Telitacicept (Active Comparator): 160mg Telitacicept was subcutaneously injected to patients with systemic lupus erythematosus at the outer side of upper arm every week for 24 weeks.
  Interventions: Drug: Telitacicept
- low dose IL2 (Active Comparator): Interleukine-2 was first added to the original treatment for systemic lupus erythematosus with 1 million IU qod for 12 weeks, injected subcutaneously at the outer side of upper arm, abdomen and thigh, then the same dose of IL2 was injected once a week for 12 weeks subcutaneously.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Telitacicept — 160mg Telitacicept was subcutaneously injected to patients with systemic lupus erythematosus at the outer side of upper arm every week for 24 weeks.
  Other Names: RC-18
  Arms: Telitacicept; Telitacicept and low dose IL2
Drug: Interleukin-2 — Low lose interleukine-2 at a dose of 1 million IU was injected once every other day for 12 weeks, then the same dose of IL2 was injected once a week at the second stage for 12 weeks.
  Other Names: Recombinant Human interleukine-2
  Arms: Telitacicept and low dose IL2; low dose IL2

SUMMARY:
The purpose of this study was to explore the clinical and immunological efficacy of Telitacicept and low dose IL-2 on systemic lupus erythematosus.

DETAILED DESCRIPTION:
Given that Telitacicept and low dose IL2 have been widespreadly applied in the treatment of systemic lupus erythematosus, this study designed a randomised, single center, prospective study to investigate the effects and safety of combined utilization of Telitacicept and low dose IL-2. 160mg Telitacicept and 1 million IU IL2 were regularly administered according to different circumstances. Then, the investigators evaluated the improvement of clinical and laboratory indexes and monitored the changes of immune cell subsets and cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at screening visits
2. Patients meet the American-European Consensus Group 2002 classification criteria of SLE.
3. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.
4. Dosing of antimalarials, prednisone or equivalent, cholinergic stimulants, and topical cyclosporine required to be stable for at least 4 weeks before screening and during study; maximum doses allowed:

   * Hydroxychloroquine, 400 mg/day;
   * Prednisone, 10 mg/day

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Laboratory abnormality: • Hb≤9 g/dl • Neutrophil 10 mg/d) within 1 month.
2. Serious complications: including heart failure (≥ New York Heart Association (NYHA) class III), renal insufficiency (creatinine clearance ≤ 30 ml/min), liver dysfunction (serum Alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of normal, or total bilirubin greater than Normal upper limit.
3. Known allergies, hyperreactivity or intolerance of tofacitinib or its excipients.
4. Have a serious infection needing hospitalization (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, EB virus, tuberculosis infection), or use intravenous antibiotics to treat infection in 2 months before the enrollment.
5. Infection with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, it is recommended to consult a doctor who has expertise in treating HIV or hepatitis C virus infection.
6. Any known history of malignancy in the past 5 years (except for nonmelanoma skin cancer, non-melanoma skin cancer or cervical tumor without recurrence within 3 months after surgical cure prior to the first study preparation).
7. Uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past 3 years, may hinder the successful completion of the study.
8. Pregnant, lactating women (WCBP) are reluctant to use medically approved contraceptives during treatment and 12 months after treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of SLE Responder Index (SRI)4 response | Week 24
  The number of participants who achieved SRI4 response at week 24.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Week 24
  The number of participants with Adverse Events throughout the study were accessed.
Autoantibody change from baseline | Week 12 and 24
  Blood samples were collected at indicated time-points for analysis of autoantibodies like anti-double stranded deoxyribonucleic Acid(dsDNA). Baseline is defined as the Day 0 visit from parent studies.
Change of complement C3 and C4 Levels from baseline | Week 12 and 24
  Blood samples were collected at indicated time-points for analysis of complement levels like complement 3 (C3) and complement 4 (C4). Baseline is defined as the Day 0 visit from parent studies.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China